CLINICAL TRIAL: NCT06144879
Title: The Biomechanics and Clinical Application of Novel Dual-headed Pedicle Screws in the Corrective Surgery for Spinal Deformity
Brief Title: Novel Pedicle Screws Used for Corrective Surgery in Spinal Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: qinxiaodong1991
Record Dates: First submitted 2023-01-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-11

CONDITIONS: Spine Deformity
Keywords: dual-headed pedicle screw

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the double-rod group (Experimental): posterior spinal corrective surgery with osteotomy (two rods without dual-headed screw)
  Interventions: Procedure: double rods without dual-headed screw
- the three-rod group (Experimental): posterior spinal corrective surgery with osteotomy (three rods with one dual-headed screw)
  Interventions: Procedure: three rods with one dual-headed screw
- the four-rod group (Experimental): posterior spinal corrective surgery with osteotomy (four rods with two dual-headed screws)
  Interventions: Procedure: four rods with two dual-headed screw

INTERVENTIONS:
Procedure: double rods without dual-headed screw — adult patients with severe spinal deformity who underwent PSO osteotomy and posterior spinal corrective surgery with traditional double rods (No dual-headed screw used)
  Arms: the double-rod group
Procedure: three rods with one dual-headed screw — adult patients with severe spinal deformity who underwent PSO osteotomy and posterior spinal corrective surgery with three rods (one dual-headed screw used in unilateral side)
  Arms: the three-rod group
Procedure: four rods with two dual-headed screw — adult patients with severe spinal deformity who underwent PSO osteotomy and posterior spinal corrective surgery with four rods (two dual-headed screw used in bilateral side)
  Arms: the four-rod group

SUMMARY:
There are still a large number of severe spinal deformity cases which would keep progressing without treatment. These patients not only have severe appearance deformity, but also suffer from cardiopulmonary compression, reduced abdominal volume, and even spinal cord injury. It is crucial to provide safe and effective surgical intervention for these patients. The corrective surgery with 3-column osteotomy is reported to be an effective surgical strategy for severe spinal deformity. However, due to the great corrective stress on the rods, there is an increased number of patients requiring revision surgery due to rod fracture (3.7%-15%). In patients with 3-column osteotomy, the osteotomy area and the upper and lower adjacent segments are mostly stress-concentrated areas, and the rod is prone to fatigue fracture. Therefore, it is necessary to reinforce the osteotomy area and adjacent segments to reduce the risk of rod fracture. Our previous study found the risk of rod fracture could be reduced by using satellite rods with duet connectors or dominos. However, in the traditional satellite rod technology, the connection of the main rod and the satellite rod rely on the traditional single slot screw and duet connectors. The two are separated and not a whole in the mechanical structure. The stability of the fixation is relatively insufficient, and stil deserves room for improvement.

Based on the traditional duet connectors, we further invent a novel dual-headed pedicle screw, which is an combination of traditional single slot screw and duet connector. Compared with the traditional duet connector, the novel dual-headed pedicle screw theoretically has stronger stability between the main rod and satellite rod, due to its integration of screw and connector. Hence, the purpose of this study is to verify the strong stability of the novel dual-headed screw by biomechanical study in cadavers performed with long spinal fusion (T12-pelvis) with L3 pedicle subtraction osteotomy (PSO). And to further investigate its effectiveness in severe adult spinal deformity patients receiving corrective surgery with PSO.

If the biomechanical properties and clinical effects of the novel dual-headed screw have been confirmed, the promotion of the product has great prospects in the world. The severe spinal deformity patients would benefit from this study when they receive spinal corrective surgery with 3-column osteotomy, using satellite rods technology by this novel dual-headed screw.

DETAILED DESCRIPTION:
Kyphosis or scoliosis is a deformity of the three-dimensional structure of the spine caused by lateral or posterior displacement of the spine. According to the population incidence statistics, the number of patients with spinal deformity in China is more than 3 million. The continuous progression of untreated or improper spinal deformity not only causes severe deformity, but also compresses the heart, lung, neurospinal cord and other important organs, leading to cardiopulmonary failure, paraplegia and even death, bringing huge economic and social burden to the country and society.

Conventional spinal orthosis uses common pedicle screws and rods to straighten the twisted spine by turning the rods and pushing and pulling screws (multiple screws one rod mode). Compared with developed countries, there are a large number of patients with moderate to severe spinal deformity in China, and there are many problems in conventional orthopaedic techniques :(1) severe spinal deformity stiffness, often requiring three-column osteotomy, spinal cord distortion and shearing during orthopaedic and closure, and the incidence of neurological complications significantly increased (8%-23%); (2) The stress between screws and rods is concentrated, and the risk of fracture after traditional internal fixation is higher (5%-22%); (3) Complex spinal malformations (such as lumbosacral or cervix and chest malformations), the installation of orthopedic rod is difficult, time-consuming and laborious operation. Therefore, it is necessary to invent new orthopaedic internal fixation devices and techniques for the safe and effective treatment of numerous patients with moderate and severe complex spinal deformity in China.

The development of three-dimensional orthopaedic theory of spinal deformity and the application of three-column spinal osteotomy have significantly improved the surgical efficacy of severe spinal deformity. In recent years, the most widely used three-column spinal osteotomy mainly includes pedicle subtraction osteotomy (PSO) and total vertebral column osteotomy (VCR), both of which can achieve good effect. The correction rate was about 50%-70% . However, with the wide development of three-column spinal osteotomy and orthopaedic surgery, the number of patients needing revision surgery due to the complications of internal fixation failure such as broken rod is increasing. Previous literature reported that the complication rate of broken rod after severe spinal deformity was about 3.7%-15%. Suk et al. reported that the incidence of rod breakage after posterior VCR for severe spinal deformity was 7.1% (5/70). Smith et al. reported that the incidence of broken rod after PSO in adult spinal deformity patients was 15.8%. Lv et al. discussed the risk factors and management strategies of rod breakage after posterior VCR surgery for severe spinal deformity, and found that the incidence of rod breakage after surgery was 3.7%. Wang Fei et al. retrospectively analyzed 7 patients with rod breakage after posterior VCR, and found that rod breakage occurred mostly within 2 years after surgery, and residual kyphosis was an important risk factor for rod breakage after surgery. Other risk factors included trauma, anterior column defect, swing gait, single rod fixation and titanium mesh displacement, etc. In patients with tri-column spinal osteotomy, the osteotomy area and adjacent upper and lower segments are mostly stress concentrated areas, and the stable osseous fusion has not been formed in the short term after surgery, and the internal fixation rod is prone to fatigue fracture. Therefore, reinforcement of the osteotomy area and adjacent segments is required to reduce the risk of rod fracture. In the past, in order to reduce the occurrence of postoperative complications of rod breakage, the commonly used improvement methods mainly include anterior support, increasing implant density and using thick rods. Anterior titanium mesh support has disadvantages such as difficulty in placement and postoperative subsidence, while increasing implant density and using thick rods will increase the cost of patients, and still cannot completely avoid the occurrence of postoperative rod breakage.

In the international scoliosis surgical orthosis mode, a long rod on the left and right sides of the spine is generally inserted into a single slot screw internal locking fixation. However, a major feature of severe scoliosis is the severe imbalance of the spine and the stiffness of the malformed segment, which makes the above traditional orthopaedic model difficult to achieve. Currently, scholars have widely recognized that the use of satellite rod technology in the periosteotomy area can reduce the risk of postoperative internal fixation failure in spinal deformity orthopaedic surgery. Scheer et al. showed in vitro biomechanical results that, compared with posterior internal fixation alone, the application of satellite rod technology in the peripherally fractured rod area could restore spinal strength during flexion, extension and left-right rotation, and the position of satellite rod was independent of spinal strength after revision. In 2012, the applicant team took the lead in applying the satellite rod technology in the three-column osteotomy for severe spinal deformity in China. The pedicle screws in the upper and lower segments of the osteotomy area were replaced by double-headed screws, making the screw placement simple. In addition, this technique does not increase the implant density of pedicle screws, and the satellite rods are mostly cut short rods, so there is no additional cost for patients. Relevant research results have been published in Spine and Chinese Journal of Orthopedics, etc.

However, in the traditional satellite rod technology, the fixation and connection of the main rod and the satellite rod rely on the traditional single slot screw and the traditional double slot connector, which are separated and not a whole in the mechanical structure, the stability of the rod is relatively poor, and the stability of the screw is insufficient. Applicants team early in order to solve the clinical problem, invented a kind of brand-new monomers double groove pedicle screws and internal fixation device, the new screw is always screw, on the basis of the traditional single slot screws and double groove connector combinations, constructed a new kind of monomers double groove pedicle screws (hereinafter referred to as new type double screw). The double-headed nail comprises a fixed end and a connecting end, and the connecting end is provided with two connecting slots: the main connecting slot and the auxiliary connecting slot. During the middle and posterior column osteotomy, double-headed nails were implanted at the head and tail of the osteotomy area, and satellite rods were placed across the osteotomy area and locked in the auxiliary connecting groove to keep the osteotomy area in a stable state during the osteotomy process. Then, the osteotomy point was closed by adjusting the satellite rods, and the main fixation rod was finally assembled.

The purpose of this study :(1) to investigate whether the multi-rod orthopaedic technique using a new double-headed screw after PSO osteotomy can improve the range of motion and biomechanical properties of the main rod strain. (2) To explore the feasibility of applying the new double-headed screw in PSO surgery for severe spinal deformity in adults, and to evaluate whether this technique can reduce the incidence of complications such as broken rod and improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. receive spinal corrective surgery from 2015-2020
2. Age: 18-70 years old
3. the Cobb angle of scoliosis or kyphosis more than 70 °
4. posterior pedicle subtraction osteotomy(PSO), using novel duet screws in three-rod or four-rod group
5. follow-up more than 24 months

Exclusion Criteria:

1. previously received spinal surgery
2. clinical and radiographic data preoperatively, postoperatively and last follow up were incomplete

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cobb angle of scoliosis (°) | 1 week after operation
  Radiographic parameters measured on X-ray by Surgimap: the angle of the major curve in coronal X-ray
Cobb angle of kyphosis (°) | 1 week after operation
  Radiographic parameters measured on X-ray by Surgimap: the angle of the kyphosis in sagittal X-ray
Coronal balance (mm) | 1 week after operation
  Radiographic parameters measured on X-ray by Surgimap: the distance between C7 plumb line (C7PL) and center sacral vertical line (CSVL) in coronal X-ray
Sagittal balance (mm) | 1 week after operation
  Radiographic parameters measured on X-ray by Surgimap: the distance between C7PL and the posterior edge of sacrum in sagittal X-ray
Rod broken rate (%) | 1 week after operation
  The ratio: number of patients with rod broken/ number of patients received surgery
Screw broke rate(%) | 1 week after operation
  The ratio: number of patients with screw broken/ number of patients received surgery
Coronal decompensation rate(%) | 1 week after operation
  The ratio: number of patients with coronal decompensation / number of patients received surgery
Sagittal decompensation(%) | 1 week after operation
  The ratio: number of patients with sagittal decompensation / number of patients received surgery
Short form-36 health survey（SF-36） | 1 week after operation
  SF-36 were calculated, including physical functioning, role physical, bodily pain, general health, vitality,social functioning, role-emotional and mental health.The SF-36 score is expressed as a number between 0 and 100. The higher the number, the better the health outcome.
Cobb angle of scoliosis (°) | 2 years after operation
  Radiographic parameters measured on X-ray by Surgimap: the angle of the major curve in coronal X-ray
Cobb angle of kyphosis (°) | 2 years after operation
  Radiographic parameters measured on X-ray by Surgimap: the angle of the kyphosis in sagittal X-ray
Coronal balance (mm) | 2 years after operation
  Radiographic parameters measured on X-ray by Surgimap: the distance between C7PL and CSVL in coronal X-ray
Sagittal balance (mm) | 2 years after operation
  Radiographic parameters measured on X-ray by Surgimap: the distance between C7PL and the posterior edge of sacrum in sagittal X-ray
Rod broken rate (%) | 2 years after operation
  The ratio: number of patients with rod broken/ number of patients received surgery
Screw broke rate(%) | 2 years after operation
  The ratio: number of patients with screw broken/ number of patients received surgery
Coronal decompensation rate(%) | 2 years after operation
  The ratio: number of patients with coronal decompensation / number of patients received surgery
Sagittal decompensation(%) | 2 years after operation
  The ratio: number of patients with sagittal decompensation / number of patients received surgery
Short form-36 health survey（SF-36） | 2 years after operation
  SF-36 were calculated, including physical functioning, role physical, bodily pain, general health, vitality,social functioning, role-emotional and mental health.The SF-36 score is expressed as a number between 0 and 100. The higher the number, the better the health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Sha, Ph.D, Study Director — Medical Ethics Committee of Drum Tower Hospital affiliated to Nanjing University School of Medicine
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim KT, Lee SH, Suk KS, Lee JH, Jeong BO. Outcome of pedicle subtraction osteotomies for fixed sagittal imbalance of multiple etiologies: a retrospective review of 140 patients. Spine (Phila Pa 1976). 2012 Sep 1;37(19):1667-75. doi: 10.1097/BRS.0b013e3182552fd0. PMID 22433502
- [Background] Zhang Y, Hai Y, Tao L, Yang J, Zhou L, Yin P, Pan A, Zhang Y, Liu C. Posterior Multiple-Level Asymmetrical Ponte Osteotomies for Rigid Adult Idiopathic Scoliosis. World Neurosurg. 2019 Jul;127:e467-e473. doi: 10.1016/j.wneu.2019.03.173. Epub 2019 Mar 25. PMID 30922897
- [Background] Suk SI, Kim JH, Kim WJ, Lee SM, Chung ER, Nah KH. Posterior vertebral column resection for severe spinal deformities. Spine (Phila Pa 1976). 2002 Nov 1;27(21):2374-82. doi: 10.1097/00007632-200211010-00012. PMID 12438987
- [Background] Smith JS, Shaffrey CI, Ames CP, Demakakos J, Fu KM, Keshavarzi S, Li CM, Deviren V, Schwab FJ, Lafage V, Bess S; International Spine Study Group. Assessment of symptomatic rod fracture after posterior instrumented fusion for adult spinal deformity. Neurosurgery. 2012 Oct;71(4):862-7. doi: 10.1227/NEU.0b013e3182672aab. PMID 22989960
- [Background] Scheer JK, Tang JA, Deviren V, Buckley JM, Pekmezci M, McClellan RT, Ames CP. Biomechanical analysis of revision strategies for rod fracture in pedicle subtraction osteotomy. Neurosurgery. 2011 Jul;69(1):164-72; discussion 172. doi: 10.1227/NEU.0b013e31820f362a. PMID 21336218
- [Background] Zhu ZZ, Chen X, Qiu Y, Chen ZH, Li S, Xu L, Sun X. Adding Satellite Rods to Standard Two-rod Construct With the Use of Duet Screws: An Effective Technique to Improve Surgical Outcomes and Preventing Proximal Junctional Kyphosis in Posterior-Only Correction of Scheuermann Kyphosis. Spine (Phila Pa 1976). 2018 Jul 1;43(13):E758-E765. doi: 10.1097/BRS.0000000000002489. PMID 29189571
- [Derived] He Z, Chen Y, Liu Z, Yang B, Shi B, Wang Y, Feng Z, Zhang T, Chen X, Qiu Y, Qin X, Zhu Z. Biomechanical Advantages of Novel Duet Screws Plus Bilateral Satellite Rods Fixation in the Correction Surgery for Adult Spinal Deformity. Orthop Surg. 2025 Aug;17(8):2454-2466. doi: 10.1111/os.70121. Epub 2025 Jul 16. PMID 40667831